CLINICAL TRIAL: NCT06060951
Title: To Investigate the Relationship Between Estimated Intraperitoneal Pressure and Non-infectious Peritoneal Dialysis (PD)-Related Abdominal Complications
Brief Title: Relating Abdominal Complications With Peritoneal Pressure Estimation and Reporting
Acronym: RAPPER
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 23HH8380; 326995 (Other: IRAS)
Record Dates: First submitted 2023-09-21; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Peritoneal Dialysis; Kidney Failure, Chronic; Hernia, Abdominal
Keywords: Intraperitoneal pressure; Gastrointestinal complications; pleuroperitoneal fistulas; patent processus vaginalis; hernia
MeSH Terms: conditions — Kidney Failure, Chronic; Hernia, Abdominal; Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Incident cohort: Including all patients from the time of PD catheter insertion until 8 weeks after starting PD
  Interventions: Diagnostic Test: Estimated intraperitoneal pressure
- Prevalent cohort: Including all patients treated with PD who are greater than 8 weeks from the start of dialysis.
  Interventions: Diagnostic Test: Estimated intraperitoneal pressure

INTERVENTIONS:
Diagnostic Test: Estimated intraperitoneal pressure — The following anthropometric measurements are required:
  1. Height: measured standing with shoes off
  2. Weight: "dry weight" should be used
  3. The distance from the decubitus plane to the mid-axillary line was measured
  4. Waist circumference: measured with a tape measure wrapped above the iliac crests around the level of the umbilicus.
  The estimated IPP will be assessed using different equations.

SUMMARY:
This is a prospective observational study in people treated with peritoneal dialysis for kidney failure to investigate whether estimated intraperitoneal pressure (eIPP) is correlated with non-infectious PD-related complications in end-stage renal failure patients. It looks to understand how both peritoneal dialysis complications (including fluid leaks and hernias) along with gastrointestinal symptoms are associated with eIPP in people treated with PD.

DETAILED DESCRIPTION:
Peritoneal dialysis is an important treatment option for kidney failure. It involves the instillation of fluid into the peritoneal cavity. The choice of volume of fluid used has a limited evidence base but will be between 1 liter to 2.5 liters depending on clinical preference. The intraperitoneal pressure (IPP) that results from this fluid varies widely between patients. However, IPP is difficult to implement clinically. There is some evidence that higher IPP is associated with an increased rate of non-infectious PD complications. These complications are mainly leaks (escape of peritoneal fluid from the peritoneal cavity) and hernias.

New methods for estimating IPP (eIPP) have been recently developed but not validated clinically. This study looks to the association of eIPP and non-infectious PD complications as well as understanding whether there is an association between eIPP and patients' burden of symptoms.

This is an observational study, no changes to fill volume or treatment will result from the eIPP. Clinicians and nurses involved in the care of the patient will not receive feedback on the eIPP measurement. This simple study will look to recruiting patients with informed consent. Those who agree to enter the study will have a small number of non-invasive measurements made at the time of a routine clinic visit. A short survey will also be administered both at the initial visit, along with 3 and 12 months later. The research team, will review the patients' notes at 12 months following recruitment for evidence of non-infectious PD-related complications.

This research proposal has informed by interaction with people with lived experience. The scientific rationale has been tested by a discussion with experts in PD in other centres.

Given that this is an observational study, individuals will not be exposed to increased clinical risk through the alteration of PD fill volume or novel procedures. The greatest burden for participants will be the completion of three short, validated survey questionnaires over 12 months.

Confidentiality will be maintained with the use of pseudonymisation to maintain participants confidentiality.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Diagnosis of end-stage renal failure requiring peritoneal dialysis as renal replacement therapy
* Ability to give informed consent and comply with study procedures.

Exclusion Criteria:

* Known allergy or hypersensitivity to any component of the dialysis solution.
* Inability or unwillingness to comply with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with kidney failure treated with peritoneal dialysis are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Non-infectious peritoneal dialysis (PD)-related complications | 3 and 12 months following study recruitment.
  Incidence of non-infectious peritoneal dialysis (PD)-related complications identified by the clinical team caring for the patient including the development of a new:
  * Hernia
  * Pleuroperitoneal fistula (PPF)
  * Patent processus vaginalis (PPV)
  * Retroperitoneal leak

SECONDARY OUTCOMES:
Gastrointestinal complications | 3 and 12 months following study recruitment.
  Patient-reported outcome changes on the Gastrointestinal Symptom Rating Scale (GSRS) questionnaire:
  GSRS is a 15-item interview-based scale, each rated on a 7-point Likert scale (1-7), higher scores indicating worse symptoms.
  GSRS items fall into five scales:
  1. Abdominal pain (includes abdominal pain, hunger pains, and nausea)
  2. Reflux syndrome (covers heartburn and acid regurgitation)
  3. Diarrhoea syndrome (encompasses diarrhoea, loose stools, and urgent need for defecation)
  4. Indigestion syndrome (includes borborygmus, abdominal distension, eructation, and increased flatus)
  5. Constipation syndrome (covers constipation, hard stools, and feeling of incomplete evacuation) Scores are calculated as the mean of completed items within each scale (min score: 1, max score: 7), higher scores indicating more severe symptoms.
  We also track the number of participants referred for surgical fixation of non-infectious PD-related complications.
Change of dialysis modality | 3 and 12 months following study recruitment.
  Number of Participants with modality change to automated peritoneal dialysis (APD) Number of Participants with transferring to haemodialysis due to non-infectious complications

CONTACTS AND LOCATIONS:
Overall Officials: Richard Corbett, PhD, Principal Investigator — Imperial College Healthcare NHS Trust
Locations (2):
- United Kingdom (2):
  - Birmingham Heartlands Hospital, Birmingham
  - Hammersmith Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
The Chief Investigator will preserve the confidentiality of participants taking part in the study and is registered under the Data Protection Act.
  Participants' information will be pseudonymized when possible. Only the pseudonymized form of data will be shared with researchers from other organizations, such as universities, National Health Service (NHS) organizations, or companies involved in health and care research in the UK or abroad, in compliance with ethical and legal requirements.
  Data collection, storage, and analysis will comply with data protection regulations, including the UK General Data Protection Regulation (UK GDPR) and the Data Protection Act 2018. All participants' information will be stored securely and analyzed using a local computer with strict arrangements for access and use, ensuring that the information is used only for health and care research or to contact participants about future research opportunities. No cloud service will be involved.
Supporting Information: Study Protocol, ICF
Time Frame: Patients' personal data will be stored in the local electronic patient management system as this is part of their follow- up and clinical care. Results of descriptive statistics or data analysis will be stored for 5 years.
Access Criteria: Only the pseudonymized form of data will be shared with researchers from other organizations, such as universities, NHS organizations, or companies involved in health and care research in the UK or abroad, in compliance with ethical and legal requirements.

REFERENCES:
- [Background] Bello AK, Okpechi IG, Osman MA, Cho Y, Cullis B, Htay H, Jha V, Makusidi MA, McCulloch M, Shah N, Wainstein M, Johnson DW. Epidemiology of peritoneal dialysis outcomes. Nat Rev Nephrol. 2022 Dec;18(12):779-793. doi: 10.1038/s41581-022-00623-7. Epub 2022 Sep 16. PMID 36114414
- [Background] Leblanc M, Ouimet D, Pichette V. Dialysate leaks in peritoneal dialysis. Semin Dial. 2001 Jan-Feb;14(1):50-4. doi: 10.1046/j.1525-139x.2001.00014.x. PMID 11208040
- [Background] Chan R, Walker RJ, Samaranayaka A, Schollum J. Long-term impact of early non-infectious complications at the initiation of peritoneal dialysis. Perit Dial Int. 2023 Jan;43(1):53-63. doi: 10.1177/08968608221132647. Epub 2022 Nov 3. PMID 36325812
- [Background] Outerelo MC, Gouveia R, Teixeira e Costa F, Ramos A. Intraperitoneal pressure has a prognostic impact on peritoneal dialysis patients. Perit Dial Int. 2014 Sep-Oct;34(6):652-4. doi: 10.3747/pdi.2012.00192. No abstract available. PMID 25228214
- [Background] Fischbach M, Terzic J, Becmeur F, Lahlou A, Desprez P, Battouche D, Geisert J. Relationship between intraperitoneal hydrostatic pressure and dialysate volume in children on PD. Adv Perit Dial. 1996;12:330-4. PMID 8865930
- [Background] Fischbach M, Desprez P, Donnars F, Geisert J. Hydrostatic intraperitoneal pressure in children on peritoneal dialysis: practical implications. An 18-month clinical experience. Adv Perit Dial. 1994;10:294-6. PMID 7999848
- [Background] Castellanos LB, Clemente EP, Cabanas CB, Parra DM, Contador MB, Morera JCO, Daly JA. Clinical Relevance of Intraperitoneal Pressure in Peritoneal Dialysis Patients. Perit Dial Int. 2017 Sep-Oct;37(5):562-567. doi: 10.3747/pdi.2016.00267. Epub 2017 Jul 11. PMID 28698250
- [Background] Scanziani R, Dozio B, Baragetti I, Maroni S. Intraperitoneal hydrostatic pressure and flow characteristics of peritoneal catheters in automated peritoneal dialysis. Nephrol Dial Transplant. 2003 Nov;18(11):2391-8. doi: 10.1093/ndt/gfg353. PMID 14551372
- [Background] de Jesus Ventura M, Amato D, Correa-Rotter R, Paniagua R. Relationship between fill volume, intraperitoneal pressure, body size, and subjective discomfort perception in CAPD patients. Mexican Nephrology Collaborative Study Group. Perit Dial Int. 2000 Mar-Apr;20(2):188-93. PMID 10809242
- [Background] Li X, Ma T, Hao J, Song D, Wang H, Liu T, Zhang Y, Abi N, Xu X, Zhang M, Sun W, Li X, Dong J. Novel equations for estimating intraperitoneal pressure among peritoneal dialysis patients. Clin Kidney J. 2023 Feb 2;16(9):1447-1456. doi: 10.1093/ckj/sfad021. eCollection 2023 Sep. PMID 37664572
- [Background] Dejardin A, Robert A, Goffin E. Intraperitoneal pressure in PD patients: relationship to intraperitoneal volume, body size and PD-related complications. Nephrol Dial Transplant. 2007 May;22(5):1437-44. doi: 10.1093/ndt/gfl745. Epub 2007 Feb 17. PMID 17308323
- [Background] Yi C, Wang X, Ye H, Lin J, Yang X. Patient-reported gastrointestinal symptoms in patients with peritoneal dialysis: the prevalence, influence factors and association with quality of life. BMC Nephrol. 2022 Mar 9;23(1):99. doi: 10.1186/s12882-022-02723-9. PMID 35264119
- [Background] Durand PY, Chanliau J, Gamberoni J, Hestin D, Kessler M. Routine measurement of hydrostatic intraperitoneal pressure. Adv Perit Dial. 1992;8:108-12. PMID 1361762
- [Background] Schmitt CP, Zaloszyc A, Schaefer B, Fischbach M. Peritoneal dialysis tailored to pediatric needs. Int J Nephrol. 2011;2011:940267. doi: 10.4061/2011/940267. Epub 2011 Jun 8. PMID 21761001
- [Background] Du BOIS D, Du BOIS EF. CLINICAL CALORIMETRY: TENTH PAPER A FORMULA TO ESTIMATE THE APPROXIMATE SURFACE AREA IF HEIGHT AND WEIGHT BE KNOWN. Archives of Internal Medicine. 1916;XVII(6_2): 863-871. https://doi.org/10.1001/archinte.1916.00080130010002

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-21): https://cdn.clinicaltrials.gov/large-docs/51/NCT06060951/Prot_SAP_000.pdf
  • Informed Consent Form (2023-09-11): https://cdn.clinicaltrials.gov/large-docs/51/NCT06060951/ICF_001.pdf